CLINICAL TRIAL: NCT06766188
Title: Online Video Training for Teachers to Improve Reading Skills in Children Using Augmentative and Alternative Communication
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold University College (Other)
Collaborators: University of South-Eastern Norway (Other); Federal University of São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 689536; 344349 (Other Grant/Funding Number: The Research Council of Norway)
Record Dates: First submitted 2024-11-29; First posted 2025-01-09 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Autism; Intellectual Disabilities
Keywords: intellectual disabilities; AAC; Shared reading; reading intervention; Sound blending; letter-sound correspondence; Phoneme segmentation; Decoding; sight words; education; online video training
MeSH Terms: conditions — Autistic Disorder; Intellectual Disability | interventions — Proto-Oncogene Proteins c-raf

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video training for teachers (Active Comparator): It is 14 schools and they will be randomized into two groups. The teachers at seven schools will receive video training on how to carry out the reading intervention.
  Interventions: Other: Online Video training for Teachers based on Reading for all
- In-person mentoring for teachers (Experimental): It is 14 schools and they will be randomized into two groups. The teachers at seven schools will receive in-person training on how to carry out the reading intervention
  Interventions: Other: Online Video training for Teachers based on Reading for all

INTERVENTIONS:
Other: Online Video training for Teachers based on Reading for all — Reading intervention over a year for students with intellectual disabilities who use AAC. This study included teachers from 14 different schools and 8 municipalities and their students. It is two arms in the intervention, with approximately 7 schools and their teachers in "video training for teachers" and "in person mentoring for teachers". The schools are randomized into these two groups, but in both groups, they will carry out the same intervention.
  The students in both groups will work explicitly and systematically with the reading material "Reading for all", which is based on the research of, among others, Janice Light and David McNaughton, and their reading program "Accessible Literacy Learning (ALL)".

SUMMARY:
The aim of this study is to investigate , via a randomized control trial (RCT), the effectiveness of an online video training platform designed for teachers to support the improvement of basic reading skills of children with intellectual disabilities (ID) who require augmentative and alternative communication (AAC). This intervention will include 14 schools and 70 students with ID who require AAC age 6-14 years old. The research question is:

1) What is the difference between online video training and in-person training on improving word-level readig skills and phonological awareness?

The students will work with a reading material, Reading for All, that follow the strategies of Accessible Literacy Learning, developed by Janice Light and David McNaughton. Reading for All is based on the research of Janice Light and David McNaughton. The reading material are adapted for AAC-users and the students can answer with pointing or their AAC-systems. Teachers will implement the instructions at the students familiar place at school for three to five days, each week, for a year.

The reading material consist of tasks in sound blending, letter-sound correspondence, phoneme segmentation, sight words, shared reading and decoding. The teachers will use evidence based, systematic and explicit instructions and immediate and corrective feedback

DETAILED DESCRIPTION:
Children with disabilities who require AAC may experiance challenges in various areas development, including communication skills, speech, language, cognitive and conceptual development, literacy, social participation, access to education, and overall quality of lifte. Acquiring reading skills may lead to higher levels of communication. Students who require AAC may be more dependent on others to provide and teach symbols to represent their language. Acquireing reading skills, may incrace the possibility to independently express themselves, and increace their access to for example text based communication devices.

There is a laci of evidence-based reading material adapted for students with ID who require AAC.

Primary outcomes will be assessed six times every two months over one year. The reading test are based on the reading material, which will be validated before the beginning of the trial.

Secondary outcome: four-time points (baseline, fourth, eighth, and twelfth month).

ELIGIBILITY:
Inclusion Criteria:

* ages 6-14 years,
* diagnosed with intellectual disability, confirmed by multidisciplinary assessments carried out by the Child rehabilitation service,
* not have a functional speech, i.e. require AAC to understand and make oneself understood,
* must use AAC as their primary form of communication,
* cannot follow ordinary curricula (LK20) but have their own education plan.

Exclusion Criteria:

* having a severe visual impairment and not being able to decode single words (e.g., severe hearing impairment).

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-03-17 (Estimated); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
Early reading skills outcome | From intervention start to the end of intervention at twelve months
  Primary outcome will be assessed six times every two months over one year.
  * Sound blending [score ranging from 0 to 15] involves testing the student's ability to combine individual sounds into words.
  * Letter-sound correspondence [score ranging from 0 to 25] involves testing the students' ability to correspond between the sounds of speech (phonemes) and the written letters representing speech (graphemes).
  * Phoneme segmentation [score ranging from 0 to 20] tests students' ability to segment the first phoneme of the word (e.g., s for sun).

SECONDARY OUTCOMES:
Reading outcome | From intervention start to the end of intervention at twelve months
  The Secondary Outcome: four-time points (baseline, fourth, eighth, and twelfth month).
  * Recognition of sight words [score ranging from 0 to 20] measures the student's ability to recognize words learned by sight.
  * Decoding [score ranging from 0 to 20] evaluates students' ability to recognize the letters in the word, associate each letter with its corresponding sound, hold these sounds in sequence in working memory, blend the sounds to determine the word, retrieve the meaning of the word.
Vocabulary | From intervention start to the end of intervention at twelve months
  The teachers will map the students communicative competance by using MacArthur-Bates Communicative Development Inventories (MCDI before and after the reading intervention to measure development of vocabulary. Score range for word and gestures have 391 words and word and sentences have 731 words.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Cogo Moreira, Professor, Principal Investigator — Ostfold University College
Locations (1):
- Østfold University College, Halden, Norway

IPD SHARING:
Plan to Share IPD: Yes
Following the FAIR Data Principles, the trial protocol, its registration, and models created to analyze the data during the project will be made available on platforms such as OSF and https://clinicaltrials.gov/. Project objectives and results will be communicated to the general public through newsletters, social media, mainstream media (regional newspaper), and presentations at showcase events. Lastly, we plan to launch a publicly accessible website of the project, describing the project, including its goals and the partners.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Study protocol: January 2025- August 2027 Statistical analysis Plan: May 2026- August 2027 Analytic Code: June 2026- August 2027

REFERENCES:
- [Background] Ulriksen LB, Bilet-Mossige M, Cogo-Moreira H, Oien R, Nordahl-Hansen A. Reading instruction for students with intellectual disabilities who require augmentative and alternative communication: A multiple single case study with baseline, posttest, follow-up, and maintenance. Res Dev Disabil. 2024 Aug;151:104790. doi: 10.1016/j.ridd.2024.104790. Epub 2024 Jun 26. PMID 38935986
- [Background] Ulriksen LB, Bilet-Mossige M, Moreira HC, Larsen K, Nordahl-Hansen A. Reading intervention for students with intellectual disabilities without functional speech who require augmentative and alternative communication: a multiple single-case design with four randomized baselines. Trials. 2023 Jun 27;24(1):433. doi: 10.1186/s13063-023-07452-4. PMID 37370125